CLINICAL TRIAL: NCT01894360
Title: A Randomized, Parallel-Group, Open-Label Study to Estimate the Relative Bioavailability, Tolerability and Safety of a Single Dose of Belimumab Administered Subcutaneously to Healthy Subjects by Prefilled Syringe or Autoinjector
Brief Title: A Study to Estimate the Relative Bioavailability, Tolerability and Safety of a Single Dose of Belimumab Self-Administered Subcutaneously (SC) by Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117100
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Pharmacokinetics; Phase 1; Healthy Subjects; Comparability; Belimumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belimumab 200 mg/mL, prefilled syringe (Experimental): Subjects will be randomly assigned in a 1 to 1 ratio to receive a single dose of 200 mg belimumab SC (1.0 mL injection) via prefilled syringe on Day 0.
  Interventions: Drug: Belimumab 200 mg/mL
- Belimumab 200 mg/mL, Autoinjector (Experimental): Subjects will be randomly assigned in a 1 to 1 ratio to receive a single dose of 200 mg belimumab SC (1.0 mL injection) via prefilled syringe contained within an autoinjector device on Day 0.
  Interventions: Drug: Belimumab 200 mg/mL

INTERVENTIONS:
Drug: Belimumab 200 mg/mL — Clear to opalescent, colorless to pale yellow sterile solution sterile solution for SC injection in a single-use liquid formulation of Belimumab 200 mg/mL will be supplied in 1mL long glass prefilled syringe or autoinjector device.

SUMMARY:
This will be a randomized, parallel-group, open-label, single-dose study of belimumab in healthy subjects to estimate the relative bioavailability, tolerability and safety of a single dose of belimumab 200 milligram (mg) when self-administered SC by healthy subjects using a prefilled syringe or autoinjector. This study will also assess the usability and reliability of the injection devices. A total of approximately 80 subjects (40 per group) will be randomly assigned in a 1 to 1 ratio to receive 200 mg belimumab SC as a single 1.0 milliliter (mL) injection of the liquid formulation (200 mg/mL) on Day 0 via the assigned injection device. Subjects will continue to be followed for 70 days after the administration of belimumab.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied, may be included only if the Investigator in consultation with the GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Negative urine drug screen; A negative urine drug screen for ethanol, opioids, barbiturates, cocaine, and amphetamines is required during screening
* Body weight >=45 kilograms (kg) to 120 kg (inclusive) at Screening
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy (for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records); or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] >40 milli international units/milliliter (MlU/ml) and estradiol <40 picogram/milliliter (pg/ml) (<147 picomol/liter [pmol/L]) is confirmatory). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method; Child-bearing potential with negative pregnancy test as determined by serum or urine human chorionic gonadotropins (hCG) test at screening or prior to dosing and Agrees to use one of the contraception methods for 2 weeks prior to the day of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until Day 112, or; OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Alanine aminotransferase (ALT), alkaline phosphatase (ALP) and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged corrected QT interval (QTc) values of triplicate electrocardiograms (ECGs) obtained over a brief recording period: QTc <450 milliseconds (msec), QTc <480 msec in subjects with bundle branch block.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The use of any concomitant prescription medications within the 30 days prior to Day 0, or anticipated use during the study period. Subjects taking prescription contraceptives, HRT, over the counter medications (e.g., antihistamines), or nutritional support (vitamins, minerals, or amino acids) may be enrolled.
* Have received a live vaccine within 30 days of Day 0 or anticipate receipt of a live vaccine during the study or within 120 days after last injection of study drug.
* History of major organ transplant: e.g., heart, lung, kidney, liver, or hematopoietic stem cell transplant.
* History of malignant neoplasm within the last 5 years, except for adequately treated basal or squamous cell cancers of the skin, or carcinoma in situ of the uterine cervix.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: For UK sites: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits. For US sites: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of atopy or anaphylactic reaction to any food, drug, or insect bite/sting.
* History of allergic reaction to parenteral administration of contrast agents, foreign proteins, or monoclonal antibodies.
* History of any infection requiring hospitalization, antivirals, or antibiotics within 4 weeks prior to Day 0.
* History of or positive test for human immunodeficiency virus (HIV) at Screening.
* Grade 3 or 4 lymphopenia at Screening.
* A positive pre-study Hepatitis B surface antigen, or Hepatitis B core antibody or positive Hepatitis C antibody result within 3 months of screening.
* Grade 3/4 immunoglobulin G (IgG) deficiency and immunoglobulin A (IgA) deficiency at Screening.
* Participated in a clinical trial (ie, received the last dose) of an investigational agent within 30 days prior to screening or 5 half-lives of the drug (whichever is longer), or continues to show evidence of toxicity from an investigational agent taken during a clinical trial.
* Exposure to more than four new chemical entities within 12 months prior to Day 0.
* Received treatment with any B cell targeted therapy (eg, rituximab, other anti-CD20 agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], BLyS-receptor fusion protein [BR3], TACI-Fc, LY2127399 [anti-BAFF], belimumab or any other B cell depletor) at any time in the past.
* Is unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access to veins.
* Donated blood or have had a significant blood loss (volume ≥ 500 mL) within 56 days prior to screening. Donated plasma within 7 days prior to screening.
* Lactating females.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2014-05-13 (Actual); Study Completion 2014-05-13 (Actual)

PRIMARY OUTCOMES:
Plasma PK assessment for Cmax, AUC(0-t), AUC(0-inf) | From Baseline upto Day 70
  Blood sample will be collected for estimation of relative bioavailability and assessment of PK parameters including maximum observed concentration; Cmax, area under the concentration-time curve from time 0 to time t; AUC(0-t) and area under the concentration-time curve from time 0 to infinity; AUC(0-inf)

SECONDARY OUTCOMES:
Safety and tolerability assessment including Adverse events (AEs), serious adverse events (SAEs), changes in laboratory values, and vital signs | From Screening upto Day 70
  Safety measurements will be assessed for AEs and SAEs, clinical laboratory parameters including Clinical hematology, chemistry, serum immunoglobulin isotypes and urinalysis. Vital signs measurements including temperature, systolic and diastolic blood pressure, pulse rate and respiratory rate.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 117100 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/117100?search=study&search_terms=117100#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 117100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register